CLINICAL TRIAL: NCT02647996
Title: Functional Connectivity Measurement After Severe Traumatic Brain Injury
Acronym: Connectivite
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01873-44
Record Dates: First submitted 2015-02-26; First posted 2016-01-06 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conscious patients: group: TBI patients awoken from comatose state with normal level of consciousness.
  intervention: fMRI (resting state) and structural (DTI)
  Interventions: Procedure: MRI: functional (resting state) and structural (DTI)
- DOC patients: group: TBI patients awoken from comatose state with abnormal level of consciousness
  intervention: fMRI (resting state) and structural (DTI)
  Interventions: Procedure: MRI: functional (resting state) and structural (DTI)

INTERVENTIONS:
Procedure: MRI: functional (resting state) and structural (DTI) — One hour brain MRI recording without active task for the patient, no sedation

SUMMARY:
To compare functional connectivity after severe traumatic brain injury (TBI) between a group of post-comatose TBI with restored consciousness and a group of post-comatose TBI with persistant disorder of consciousness at admission in rehabilitation

DETAILED DESCRIPTION:
Recovery of consciousness can be impaired in severe traumatic brain injury (TBI). Prognostic factors are sparse and mostly clinical (mainly the initial Glasgow coma scale GCS) (1). Functional magnetic resonance imaging (fMRI) could allow a better understanding of functional recovery. Graph method has been applied to fMRI signal analysis in disorder of consciousness (DOC) due to post-anoxic encephalopathy. Comatose state was characterized by dramatic change in local connectivity (hub location) without significant change in global connectivity (2). The present study aims at describing functional connectivity in DOC following severe TBI. We will record resting state fMRI in TBI patients in two clinical conditions: conscious state versus DOC state.

ELIGIBILITY:
Inclusion Criteria:

* severe TBI
* no general anesthesia since 7 days
* no neuroleptic nor hypnotic drug since 3 days
* medical criteria fulfilled to be discharged from ICU
* medical insurance

Exclusion Criteria:

* age < 18
* contra indication to MRI
* consent refusal from the family
* neurological trouble before TBI
* patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe TBI admitted in ICU and ready to be discharged to rehabilitation with or without DOC
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
cortical functional connectivity | connectivity index measured on MRI recorded at discharge from intensive care unit (ICU) (30 days post-TBI on average) and compared between the two groups of patients (group "normal level of consciousness" versus group "disorder of consciousness")
  the index is calculated from methodology of the article cited below (2)

SECONDARY OUTCOMES:
consciousness level measured with Coma recovery scale -revised (CRS-R) | CRS-R score at discharge from intensive care unit (ICU) (30 days post-TBI on average)
consciousness level measured with Coma recovery scale -revised (CRS-R) | day 60 after first MRI
cortical functional connectivity change | connectivity index change (measured on MRI done day 60 after first MRI and compared to MRI done on day 0
Slow wave sleep quantification | EEG at discharge from intensive care unit (ICU) (30 days post-TBI on average)
  Electroencephalographic recording on 12 consecutive hours by night
structural connectivity | DTI At discharge from intensive care unit (ICU) (30 days post-TBI on average)
  fibers density between region of interest by DTI
structural connectivity | DTI day 60 after first MRI
  fibers density between region of interest by DTI

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Oujamaa, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

REFERENCES:
- [Background] Nakase-Richardson R, Whyte J, Giacino JT, Pavawalla S, Barnett SD, Yablon SA, Sherer M, Kalmar K, Hammond FM, Greenwald B, Horn LJ, Seel R, McCarthy M, Tran J, Walker WC. Longitudinal outcome of patients with disordered consciousness in the NIDRR TBI Model Systems Programs. J Neurotrauma. 2012 Jan 1;29(1):59-65. doi: 10.1089/neu.2011.1829. Epub 2011 Aug 4. PMID 21663544
- [Background] Achard S, Delon-Martin C, Vertes PE, Renard F, Schenck M, Schneider F, Heinrich C, Kremer S, Bullmore ET. Hubs of brain functional networks are radically reorganized in comatose patients. Proc Natl Acad Sci U S A. 2012 Dec 11;109(50):20608-13. doi: 10.1073/pnas.1208933109. Epub 2012 Nov 26. PMID 23185007